CLINICAL TRIAL: NCT05259267
Title: Investigation of the Effectiveness of an Online Group Therapy Program for Post-Traumatic Growth in Women With Breast Cancer
Brief Title: Online Group Therapy for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Cennet Yastıbaş, Research Assistant, PhD candidate, clinical psychologist, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121K686
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; post-traumatic growth; online group therapy; online support groups
MeSH Terms: conditions — Breast Neoplasms | interventions — Teniposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Group Therapy for PTG (Experimental): It consists of eight sessions that occur during app. 90 minutes. A group therapist and a cotherapist will lead the therapy sessions. There will be one session per a week.
  Interventions: Behavioral: Online Group Therapy for PTG
- Online Support Group (Active Comparator): It consists of eight sessions that occur during app. 90 minutes. A group therapist and a cotherapist will lead the therapy sessions without using any psychological methods. There will be one session per a week.
  Interventions: Behavioral: Online Support Group
- Wait-list (No Intervention): We used a wait-list as a control group. After each participants in both online PTG group therapy and online support group completed the interventions, wait-list will be randomly assigned to one of these two interventions.

INTERVENTIONS:
Behavioral: Online Group Therapy for PTG — Online Group Therapy for PTG consists of eight sessions. Each sessions have specific themes. First session: psychoeducation, normalization of the experiences and emotions. Second session: emotion regulation skills. Third session: awareness of the negative thoughts that make patients worried, anxious, feared. Forth session: restructuring of the thoughts and practicing mindfulness technics. 5. session: practicing of self-disclosure skills 6. session: creating a breast cancer story with balancing losses and gains. 7. session: sharing of the effects of breast cancer on life and developing new life priorities 8. session: making life meaning and developing new life goals.
  Arms: Online Group Therapy for PTG
Behavioral: Online Support Group — Online support groups also consist of eight sessions. 1. session: introducing the program and learning the expectancies 2. session: sharing what is known about breast cancer 3. session: risk and protective factors for breast cancer 4. session: sharing side effects of surgical operation and treatments 5. session: sharing the reactions of family, close friends 6. session: patient-doctor relationship and also sharing the challenges and facilitators of healthcare system 7. session: sharing the current position in the treatment and of what has been done for improvement 8. session: sharing the reliable information sources for breast cancer and close
  Arms: Online Support Group

SUMMARY:
Breast cancer is a serious and life-threatening health problem that is increasing all over the world and in Turkey. Although the survival rate increases with the improvement of the diagnosis and treatment processes for breast cancer, cancer patients experience some psychosocial problems both due to their treatment and the disease. Decreases in quality of life, psychological distress, especially depression and anxiety, post-traumatic stress disorder as well as sleep disorders, fatigue, fear of cancer recurrence could be common negative outcomes that experienced by the breast cancer patients. Although, cancer could be such a life-threatening disease, some patients report that they experience positive changes in their lives after the diagnosis of cancer. The concept of Post-Traumatic Growth (PTG) was first developed by Tedeschi and Calhoun (1995). PTG is a concept that refers positive psychological changes after struggling an stressful life event. According to the Functional-Descriptive model of Tedeschi and Calhoun, post-traumatic growth occurs in five areas; relating to others, personal strength, spiritual changes and appreciation of life. In this context, a group intervention program has been developed for PTG, which will bring the person to a better functionality than before the trauma to enhance the Post-Traumatic Growth level of women with breast cancer. The current research project will consist of three arms; therapy group, support group and wait-list. Online group therapy consists of eight sessions that continue approximately 90 minutes. In addition to an active treatment group for PTG, an online support group has been developed by the researchers to investigate the effectiveness of the therapy. Online support group also consists of eight sessions during approximately 90 minutes as in intervention program. Wait-list is considered as a control group. A set of reliable and validated measurement tools will be administered and heart rate variability as a physical measurement will be used to examine the effects of the therapy. The research hypotheses are based on that patients who participated active treatment group will have better PTG level and other related concept with PTG (like higher score of deliberate rumination) and better Heart-Rate Variability scores than other groups. The researcher will plan to take three time measurement: pre-intervention, post-intervention, and 1-month follw-up.

DETAILED DESCRIPTION:
Preliminary studies to development of the programs Before the development of protocol of the current treatment programs, the investigators reviewed related literature and published a systematic review about the related factors for PTG in women with breast cancer. After obtaining the ethical approval the study coordinator interviewed with eight women via telephone to explore the experiences of women with breast cancer. The investigators determined the needs and possible challenges of the illness. Besides, previous similar treatment programs were examined in detail. Later, the investigator developed the study protocol with the supervisor and send the content of the treatment programs to five specialists who have MD in clinical psychology and got feedback and the investigators revisited final version of the treatment programs.

In brief, the research hypotheses are 1) both online group therapy for PTG and online support groups will show better PTG levels and rumination scores, and other secondary measurements (such as psychological distress, heart rate variability, disclosure of distress) than wait-list control. 2) Participants who in online group therapy for PTG will improve better PTG and rumination scores, and secondary measurements' scores compared with the participants in online support groups. 3) The benefits of the treatment programs will be endured for 1-month follow-up measure.

Procedure Ethical approval: This study was approved by the institutional review board of Eskisehir Osmangazi University. All study participants gave written informed consent. Announcements will be posted in various departments of the hospital to participate in the research. First of all, volunteer participants will be assessed through the phone and informed about the research process. If they agree to participate, the investigators will organize a detailed interview. In this interview one of the researchers of the study who is a psychiatrist will apply SCID to eliminate the other possible mental disorder. Patients who meet the criteria will be informed about the group and informed consent forms will be obtained. Before beginning of the treatment program, baseline measurement and ECG Holter measurement will be scheduled by the telephone. After completing baseline measurement, the participants will then be randomly allocated to one of the three groups.

The online treatment programs will be delivered to groups of 6-8 participants by a psychologist and psychiatrist (therapist and co-therapist), eight weekly online sessions. Online sessions will be delivered through an online video-conferencing software (ZOOM). Sample size is determined by g-power analysis. For three-arm randomized controlled trial we plan to recruit at least 51 participants (each group should have at least 17 participants). Before the beginning of the study, the participants will be informed about online video-conferencing platform. The investigators will send a video about the use of platform and also step by step user manual. Each participant in treatment programs should join at least six sessions. If the participants could not complete six sessions, the investigators will admit them drop-out (This information will be declared during the interviews and written informed consent). The investigators will use SPSS 23.0 Package Program for Social Sciences. The descriptive analysis will be performed for frequencies of socio-demographics and clinical information such as cancer stage, treatments. To test the hypothesis, the investigators will conduct a repeated measure ANOVA. The investigators will employ intention to treat and as treated analysis.

ELIGIBILITY:
Inclusion Criteria:

* women who have been diagnosed with breast cancer for the first and only
* women who have been diagnosed breast cancer in 2018 and later (past four years)
* stage I, II and III patients
* ability to use internet
* having a personal computer or tablet with a camera and microphone
* describing cancer as a stressful life event (using PCL-5 to assess post-traumatic stress level)

Exclusion Criteria:

* recurrence of breast cancer,
* second cancer,
* severe psychological or physical comorbidity

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We will recruit women who diagnosed breast cancer. Our sample is considered based on biological sex.
Enrollment: 51 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change in Post-traumatic Growth Inventory | Baseline measurement before the treatment programs begin (pre-intervention),post-intervention at week 8(after completing eight week intervention), and 1-month follow-up.
  The Turkish version of Post-traumatic Growth Inventory to measure PTG levels of the patients will be used. It is compromised of 21 item and scored ranging from 0 to 5. Higher scores refer higher PTG level.
Change in Event-Related Rumination Inventory (ERRI) | Baseline measurement before the treatment programs begin (pre-intervention),post-intervention at week 8 (after completing eight-week intervention), and 1-month follow-up.
  The Turkish version of Event-Related Rumination Inventory (ERRI) that is reliable and validated measure will be used to assess rumination of the breast cancer. It has 20 items and two sub-scale; intrusive and deliberate rumination. The scores are changing from 0 to 3.
PTSD Checklist for DSM-5 (PCL-5) | Baseline measurement to deciding to join the treatment programs
  It will be used to asses stressful level of breast cancer to participate the treatment programs.The 20-item self-report measure of PTSD scored from 0 to 4, and yielding a scale score range of 0-80.

SECONDARY OUTCOMES:
Change in Depression Anxiety and Stress Scale (DASS-21) | Baseline measurement before the treatment programs begin (pre-intervention),post-intervention at week 8(after completing eight week intervention), and 1-month follow-up.
  The Turkish version of Depression Anxiety and Stress Scale which is a reliable and validated study result will be used for secondary outcome. It consists of 21 items and three sub scale. Higher scores of each sub-scale sign higher distress level.
Change in Heart-Rate Variability | Baseline measurement before the treatment programs begin (pre-intervention),post-intervention at week 8(after completing eight week intervention), and 1-month follow-up.
  Holter electrocardiogram (ECG) Monitoring will be used to asses physical effects of intervention programs. It will be used 24 hour holter. A cardiologist will read the holter ECG results. Heart rate will be analyzed using the standard deviation of sequential interbeat intervals averaged over 5 min epochs (SDANN)
Change in Distress Disclosure Index | Baseline measurement before the treatment programs begin (pre-intervention),post-intervention at week 8(after completing eight week intervention), and 1-month follow-up.
  It will be used to evaluate emotional expression and repression. Our treatments may indirectly have impact on disclosure of the patients' emotions. The Turkish version of Distress Disclosure Index which has good reliability and variability scores has 12 items and rated on a five-point scale (scored 1-5). Higher scores refer higher expression of emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Cennet Yastıbaş-Kaçar, MD, Study Chair — Dokuz Eylul University
Locations (1):
- Eskişehir Osmangazi University Faculty of Medicine, Eskişehir, Turkey (Türkiye)